CLINICAL TRIAL: NCT04879303
Title: Robotic Intervention Framework for Children With Autism Spectrum Disorder to Enhance Social Engagement and Participation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Education University of Hong Kong (Other)
Responsible Party: Principal Investigator, Eva Chung Yin-han, Assistant Professor, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R1230
Record Dates: First submitted 2021-04-19; First posted 2021-05-10 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Autism Spectrum Disorder; Social Engagement; Robotic Intervention
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Robot-assisted social skill intervention (Experimental): Social robotics will be used by the instructor to conduct the social skill training activities.
  Interventions: Behavioral: Robot-assisted social skill intervention
- Human-only instruction program on social skill training (Active Comparator): The children will receive only the human-delivered social skill training.
  Interventions: Behavioral: Human-only instruction programme on social skill training
- Control (No Intervention): There will be no intervention conducted during the tested period

INTERVENTIONS:
Behavioral: Robot-assisted social skill intervention — Social robotics will be used by the instructor to teach social skills to the children with ASD for 12 weekly sessions.
  Arms: Robot-assisted social skill intervention
Behavioral: Human-only instruction programme on social skill training — The children will receive only the human-delivered training throughout the 12 sessions, with the content and sequence of activities the same as the robotic intervention group.
  Arms: Human-only instruction program on social skill training

SUMMARY:
This study will develop and test a Robotic Intervention Framework for Children with ASD in the real context. The first part of this study will focus on the identification and initial testing of core elements of effective robotic intervention programs to form a practice framework. Pat II will use a randomized control trial to test the efficacy of the robotic intervention programs that incorporated all elements of the framework. Part III will use a qualitative approach to examine the qualitative outcomes of the program with reference to the elements of the practice framework. With a framework that is built upon evidence and tested sufficiently, practice guidelines and intervention protocol will be delineated to ensure success of robotic intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of autism spectrum disorder
* aged between 5-11
* normal intelligence

Exclusion Criteria:

* with self-injurious or aggressive behavior
* with hearing or visual impairment

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The Autism Diagnostic Observation Schedule | 1 week before the intervention
  The Autism Diagnostic Observation Schedule (ADOS) is a play-based standardized protocol for observing interaction, communication, repetitive behavior and play. It has a standardized algorithm score on communication and reciprocal social interaction domains that can contribute to diagnosis and to measure change in autistic symptoms during treatment. The ADOS creates an interactive play environment in which the children's social behaviors, use of speech and gestures in social situations can be observed. It is individual-based and will take 30-45 minutes for administering.
The Autism Diagnostic Observation Schedule | 1 week after the intervention
  The Autism Diagnostic Observation Schedule (ADOS) is a play-based standardized protocol for observing interaction, communication, repetitive behavior and play. It has a standardized algorithm score on communication and reciprocal social interaction domains that can contribute to diagnosis and to measure change in autistic symptoms during treatment. The ADOS creates an interactive play environment in which the children's social behaviors, use of speech and gestures in social situations can be observed. It is individual-based and will take 30-45 minutes for administering.
Social Responsiveness Scale | 1 week before the intervention
  The Social Responsiveness Scale (SRS) is a questionnaire which is comprised of 65 items. It systematically collects information on parents' reports of their children's social awareness, cognition, communication, motivation and mannerisms.
Social Responsiveness Scale | 1 week after the intervention
  The Social Responsiveness Scale (SRS) is a questionnaire which is comprised of 65 items. It systematically collects information on parents' reports of their children's social awareness, cognition, communication, motivation and mannerisms.
The Canadian Occupational Performance Measure | 1 week before the intervention
  The Canadian Occupational Performance Measure (COPM) is a validated tool for measuring outcomes of intervention programs on activity participation. It will collect both quantitative and qualitative data. The performance score and satisfaction score on participation of activities will be collected both before and after the intervention to reveal the change of the client throughout the intervention.
The Canadian Occupational Performance Measure | 1 week after the intervention
  The Canadian Occupational Performance Measure (COPM) is a validated tool for measuring outcomes of intervention programs on activity participation. It will collect both quantitative and qualitative data. The performance score and satisfaction score on participation of activities will be collected both before and after the intervention to reveal the change of the client throughout the intervention.
Short sensory profile | 1 week before the intervention
  The Short Sensory Profile is a validated assessment tool to capture sensory processing behaviors that indicate a low or high threshold to sensory experiences resulting in interference with the performance of daily living tasks. This parent-reported measure is scored on six sensory systems and two behavioral category subscales, namely auditory processing, visual processing, taste and smell processing, body position, movement, touch processing, activity level, and social and emotional responses. Item scores can be calculated and aggregated into the seven factor scores: emotionally reactive, sensory sensitivity, low registration, sensory seeking, sensory defensiveness, oral sensory seeking, and low endurance.
Short sensory profile | 1 week after the intervention
  The Short Sensory Profile is a validated assessment tool to capture sensory processing behaviors that indicate a low or high threshold to sensory experiences resulting in interference with the performance of daily living tasks. This parent-reported measure is scored on six sensory systems and two behavioral category subscales, namely auditory processing, visual processing, taste and smell processing, body position, movement, touch processing, activity level, and social and emotional responses. Item scores can be calculated and aggregated into the seven factor scores: emotionally reactive, sensory sensitivity, low registration, sensory seeking, sensory defensiveness, oral sensory seeking, and low endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Yin-han Chung, PhD, Principal Investigator — The Education University of Hong Kong
Locations (1):
- The Education University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung EY, Kuen-Fung Sin K, Chow DH. Effectiveness of Robotic Intervention on Improving Social Development and Participation of Children with Autism Spectrum Disorder - A Randomised Controlled Trial. J Autism Dev Disord. 2025 Feb;55(2):449-456. doi: 10.1007/s10803-024-06236-2. Epub 2024 Jan 17. PMID 38231380